CLINICAL TRIAL: NCT07077291
Title: Combining Mindfulness-Based Cognitive Therapy With Escitalopram for Cognitive and Emotional Recovery in Older Adults With Treatment-Resistant Depression
Brief Title: MBCT and Escitalopram for Treatment-Resistant Depression in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yun Zhang (Other)
Responsible Party: Sponsor-Investigator, Yun Zhang, Principal investigator, Tangshan Gongren Hospital
Organization: Tangshan Gongren Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-139
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Treatment-resistant Depression (TRD)
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: MBCT + Escitalopram Group (Experimental): Participants received mindfulness-based cognitive therapy (MBCT) in weekly 120-minute group sessions for 12 weeks, in addition to daily oral administration of escitalopram hydrobromide (20mg/day).
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy (MBCT); Drug: Escitalopram Hydrobromide
- Active Comparator: Escitalopram Alone Group (Active Comparator): Participants received daily oral administration of escitalopram hydrobromide (20mg/day) and served as the control group.
  Interventions: Drug: Escitalopram Hydrobromide

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy (MBCT) — A group intervention delivered by a psychiatrist and two assistants. Sessions were 120 minutes, once per week, for 12 weeks. Content included mindfulness exercises such as 3-minute breathing space, body scanning, mindfulness walking, meditation, and cognitive therapy techniques to observe connections between thoughts, emotions, and behavior.
  Arms: Experimental: MBCT + Escitalopram Group
Drug: Escitalopram Hydrobromide — Oral administration of escitalopram hydrobromide tablets, 20mg once daily (qd) for the entire 12-week study duration.

SUMMARY:
This study is a randomized controlled trial designed to investigate the synergistic effects of combining mindfulness-based cognitive therapy (MBCT) with escitalopram hydrobromide versus escitalopram alone on cognitive function, depressive symptoms, and quality of life in older adults diagnosed with treatment-resistant depression (TRD) and cognitive impairment.

DETAILED DESCRIPTION:
Treatment-resistant depression (TRD) in older adults presents a significant clinical challenge, often accompanied by cognitive impairment that affects daily functioning and well-being. While escitalopram is a standard pharmacological treatment, monotherapy may be insufficient for this population. Mindfulness-Based Cognitive Therapy (MBCT) has emerged as a promising psychotherapeutic intervention for depression by promoting awareness and altering negative thought patterns. This study aimed to evaluate if an integrated approach of MBCT plus escitalopram would yield superior outcomes compared to escitalopram alone. A total of 230 older adults with TRD were randomized to either a combined therapy group or a medication-only control group. Assessments of cognitive function (MoCA), depression severity (HAM-D), and quality of life (GQOLI-74) were conducted at baseline, 6 weeks, and 12 weeks to determine the efficacy of the combined intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 60 and 77 years.
* Montreal Cognitive Assessment (MoCA) scores ranging from 5 to 17.
* Diagnosis of persistent and treatment-resistant depression according to DSM-5 criteria.
* Maintained consistent use of escitalopram hydrobromide for the previous 6 months.
* Ability to independently perform daily tasks.
* Provided written informed consent and willing to adhere to study procedures and follow-up.

Exclusion Criteria:

* Primary diagnosis of schizophrenia, bipolar disorder, or other significant mental health conditions other than depression.
* Presence of advanced cancer, end-stage heart disease, or severe liver or kidney dysfunction.
* Recent history (within 12 months) of substance abuse or addiction.
* Significant visual or hearing impairments that would hinder participation.
* Participation in mindfulness therapy or similar CBT within the last year.
* Language comprehension or expression challenges precluding participation.

Ages: 60 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Function | Baseline, 6 weeks, 12 weeks
  Measured by the Montreal Cognitive Assessment (MoCA). The scale score ranges from 0-30, with higher scores indicating better cognitive function.
Change in Depression Severity | Baseline, 6 weeks, 12 weeks
  Measured by the 17-item Hamilton Depression Rating Scale (HAM-D-17). The scale score ranges from 0-52, with lower scores indicating less severe depressive symptoms.
Change in Quality of Life | Baseline, 6 weeks, 12 weeks
  Measured by the General Quality of Life Index-74 (GQOLI-74). The total score is calculated from 74 items, with higher scores indicating a better quality of life.

SECONDARY OUTCOMES:
Clinical Treatment Efficacy Rate | At 12 weeks
  Categorization of treatment effect as 'Significant', 'Effective', 'Average', or 'Ineffective' based on predefined changes in MoCA, HAM-D, and GQOLI-74 scores. The rate (%) of patients in each category was compared between groups.
Incidence of Adverse Events | Baseline, 6 weeks, 12 weeks
  Monitoring and recording of all adverse events (AEs) reported by participants or observed by clinicians throughout the study. AEs were assessed for severity and relationship to the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Tangshan Gongren Hospital, Tangshan, Hebei, China